CLINICAL TRIAL: NCT04683393
Title: A Single-centre Prospective Study to Explore the Role of Frailty in Patients With Multiple Myeloma.
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: MMM-FRAILTY16; R04443 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2020-10-22; First posted 2020-12-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples collected at baseline and throughout the study will also be stored for future studies to allow a prompt evaluation of novel biomarkers identified in the future, and therefore to accelerate the validation of these biomarkers.
  Routine blood assessments will be performed at the Manchester Royal Infirmary (MRI) laboratory as per clinical routine. Serum and leukocytes samples will be stored in multiple aliquots at -80oC to test future potential markers.
  The samples will be processed and stored at Manchester Royal Infirmary (MRI) in the laboratory of Dr Burthem. Samples will be then shipped in dry ice once a year to Glasgow to the laboratory of Prof Shiels for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: To compare the markers of frailty (MoF) in patients with multiple myeloma (MM) with the healthy subjects.
- MM Patients: Patients with multiple myeloma (MM), the aim is to assess if any of the proposed parameters and markers of frailty (e.g. biomarkers of cellular senescence and organ damage, inflammatory markers, physical tests such as gait speed and hand grip test) are associated with frailty status, defined according to the GA, at baseline.

SUMMARY:
This study aims to explore the markers of frailty in a "real world" population of MM patients, and to monitor changes to those markers throughout treatment and follow-up. Clinical, physical and biological parameters will be collected by interviewing the patients via questionnaires, physical tests and blood analyses. All these will be done during routine visits of the patients' care pathway, minimising the impact on patient lifestyles. The patients will then be stratified according to the geriatric assessment into 3 groups (fit, non-fit, frail) and the changes to these parameters will be compared within these 3 groups throughout the treatment and the follow-up phase for a minimum of 24 months. The markers of frailty will also be measured in a group of healthy subjects and the results will be compared with those of patients with MM.

The characterisation of markers of frailty will be a starting point to develop strategies to reduce the causes of frailty, hence it will reduce the treatment-related toxicity, improve quality of life and eventually the outcome for patients with MM.

DETAILED DESCRIPTION:
This project aims to characterize the markers of frailty in a population of MM patients in a "real world" setting. The clinical approach to the patients (i.e. treatment schedule, number of appointments in the hospital, invasive procedures) will not be changed compared to patients not enrolling in the study.

In particular, the primary objective of the study is:

To explore measures of frailty in MM patients: the aim is to assess if any of the proposed parameters and markers of frailty (e.g. biomarkers of cellular senescence and organ damage, inflammatory markers, physical tests such as gait speed and hand grip test) are associated with frailty status, defined according to the GA, at baseline.

The secondary objectives of the study are:

* To monitor frailty (defined by GA) and those markers of frailty (MoF) over time and evaluate treatment effects on frailty and MoF: this will explore the relationship between the markers of frailty and the tumor. Moreover, this will allow the study to assess if the frailty score at baseline is static or can be modified, in particular to observe whether frailty is improved in patients responding well to the treatment without toxicity.
* To explore the relationship of parameters and biomarkers of frailty with: treatment-related toxicity, treatment discontinuation, response to treatment, PFS and OS
* To investigate the predictive role of GA in the "real world" setting: the GA has been assessed in 3 clinical trials in more than 800 patients, but no data are available on the "real world" population where frail patients are more frequently encountered.
* To compare the MoF in patients with MM with the healthy subjects.
* To assess the relation of frailty and quality of life (QoL): in elderly and frail MM patients the QoL is one of the most important (if not the most important) objective for treatment. Investigators will investigate if the QoL perceived by the patient relates to the frailty assessment and how this varies over time.

Biological samples collected at baseline and throughout the study will also be stored for future studies to allow a prompt evaluation of novel biomarkers identified in the future, and therefore to accelerate the validation of these biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or greater
* Newly diagnosed or relapse/refractory patients with multiple myeloma including non-secretory multiple myeloma. If patients are at diagnosis, they need to have a myeloma defining events (MDE) as reported in Appendix B. If they are at relapse they need to meet the criteria for relapse as per Appendix C.
* Patients due to start any anti-myeloma treatment irrespectively from the line of treatment
* Able to provide written informed consent
* Patients enrolled in other clinical trials can be enrolled in this study. Patients will not attend the hospital more frequently if enrolled in this study. In fact all the assessment, tests and questionnaires will be done whilst the patients are attending the hospital for routine appointments.

Inclusion criteria for healthy subjects:

* Aged 50 years or greater
* Able to provide written informed consent

Exclusion Criteria:

* Not able to give informed consent
* MGUS or sMM without MDE
* Patients receiving ongoing treatment for MM with the exclusion of steroids (maximal dose of Dexamethasone 160 mg in last 2 weeks or equivalent) and radiotherapy for spinal cord compression (SCC). The reason for this exclusion is that the baseline measurements need to be done before starting a proper line of chemotherapy and not in the middle of a treatment in order to be comparable between patients.
* Patient received allogeneic stem cell transplant at any stage of treatment. The reason being that some markers (i.e. telomere length) can consistently change following an allogeneic stem cell transplant

Exclusion criteria for healthy subjects:

* Not able to give informed consent
* History of past or present cancer requiring treatment (surgery and/or radiotherapy and/or chemotherapy)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria EXPLICITLY state otherwise. Participants with the above characteristics are eligible:
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Frailty status defined according to Geriatric assessment | 18 months from Recruitment End
  Katz Activity of Daily Living (ADL) Questionnaires with a points scale of 1 or 0, with 0 dependence and 1 independence
Frailty status defined according to biomarkers of frailty: Teleomere Length | 18 months from Recruitment End
  Biomarkers: Telomere length analysis: on leukocytes and bone marrow by QPCR via the method of Cawthon
Frailty status defined according to biomarkers of frailty: miRNAs | 18 months from Recruitment End
  Biomarkers:miRNAs expression leukocytes via relative quantitative real-time PCR (qRT-PCR)
Frailty status defined according to biomarkers of frailty: CDKN2A | 18 months from Recruitment End
  Biomarkers: CDKN2A expression on leukocytes via relative quantitative real-time PCR (qRT-PCR)
Frailty status defined according to Geriatric assessment | 18 months from Recruitment End
  Lawton Instrumental Activity of Daily Living (IADL) Activities of daily living scale.Patients are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men
Frailty status defined according to Geriatric assessment | 18 months from Recruitment End
  Charlson Comorbidity Index (CCI). Predicts 10 year survival in patients with multiple comorbidities. Scale is No 0, Yes is plus score depending on disease. Lower the overall points the greater survival rate